CLINICAL TRIAL: NCT00562107
Title: Evaluation of the SafeR Mode in Patients With a Dual Chamber Pacemaker Indication
Acronym: ANSWER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANSWER - IBSY02; IBSY02
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Assess the Benefits From the AAISafeR/SafeR Algorithm of Symphony 2550 or REPLYTM DR in a Wide Range of Pacemaker Patients.
Keywords: Minimized ventricular pacing, clinical outcome, SafeR, AAIsafeR, dual chamber pacemaker therapy, % of ventricular pacing, hospitalizations, symptomatic AF

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): AAIsafeR /SafeR Patient randomized with the SafeR switched ON
  Interventions: Device: Symphony DR 2550 and REPLY DR cardiac pacemakers
- 2 (Experimental): DDD(R) mode. Patients randomized with the SafeR mode switched OFF
  Interventions: Device: Symphony DR 2550 and REPLY DR cardiac pacemakers

INTERVENTIONS:
Device: Symphony DR 2550 and REPLY DR cardiac pacemakers — AAISafeR/SafeR ON
  Arms: 1
Device: Symphony DR 2550 and REPLY DR cardiac pacemakers — DDD(R) (SafeR OFF)
  Arms: 2

SUMMARY:
The aim of this study is to assess the benefits from the AAISafeR/SafeR algorithm of Symphony 2550 or REPLY DR in a wide range of pacemaker patients.

The expected benefits will be a result of the reduction of the percentage of ventricular pacing.

It contributes to the longevity of the cardiac pacemaker and has an effect on the incidence of sustained (or persistent) Atrial Fibrillation and Heart Failure. These clinical benefits are a result of spontaneous ventricular activation which ensures a more physiological ventricular activation.

The benefits will be assessed by comparing the incidence of atrial arrhythmias and the evolution of the haemodynamic status of the patients (QOL, echo and BNP)

ELIGIBILITY:
Inclusion Criteria:

* Patient primo-implanted with a Symphony 2550 or Reply DR for less than 1 month according to the official guidelines.
* Patient implanted for sinus node dysfunction (including bradycardia-tachycardia syndrome) or 2nd, advanced or 3rd degree intermittent or allegedly permanent AV block.
* Patient implanted with a bipolar right atrial lead and a right ventricular lead
* Patient has signed a consent form after having received the appropriate information

Exclusion Criteria:

* Patient with permanent AF
* Patient suffering from sustained ventricular arrhythmias
* Patient with congenital complete heart block
* Patient with vasovagal syncope, carotid sinus syndrome
* Patient with AV node ablation
* Patient having suffered from a myocardial infarction within the last month
* Patient suffering from severe aortic stenosis
* Patient suffering from unstable angina pectoris
* Patient is not able to understand the study objectives and protocol or refuses to co-operate
* Patient is not available for scheduled follow-up
* Patient has a life expectancy less than one year
* Patient is included into another clinical study
* Patient is minor, this is < 18 years
* Patient is a pregnant woman
* Any patient with a contra-indication for the device labeling

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2007-12; Primary Completion 2011-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The outcome measure is the % of ventricular pacing and hospitalizations for specified cardiac reasons (symptomatic AF, cardioversions for AF and heart failure) | 3 years

SECONDARY OUTCOMES:
Evolution of paroxysmal AV blocks | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stockburger Martin, MD, Principal Investigator — Head of Pacemaker/Defibrillator/CRT department
Locations (37):
- 736 Cambridge Street, Brighton, Massachusetts, United States
- France (13):
  - CHU - Hopital Sud, Amiens
  - Centre hospitalier de Béthune, Béthune
  - CHU - Hopital Michallon, Grenoble
  - CHP Beauregard, Marseille
  - CHU A de Villeneuve, Montpellier
  - Clinique Bizet, Paris
  - CHU Hopital C. Nicolle, Rouen
  - CCN, Saint-Denis
  - CHU - Hopital Nord, Saint-Etienne
  - CHU Hautepierre, Strasbourg
  - Clinique Pasteur, Toulouse
  - CHU Hopital Trousseau, Tours
  - CHU de Nancy, Vandœuvre-lès-Nancy
- Germany (11):
  - Charite Virchow, Berlin
  - Bernau hospital, Bernau
  - Braunschweig hospital, Braunschweig
  - Elisabeth KH Essen, Essen
  - Leipzig Uni, Leipzig
  - Lübeck Uni, Lübeck
  - Lüdenscheid hospital, Lüdenscheid
  - Mainz Uni, Mainz
  - München Innenstadt, München
  - Remscheid hospital, Remscheid
  - Ulm Uni, Ulm
- Italy (5):
  - Clinica Villa Pini d'Abruzzo, Chieti
  - Osp Civile di Montebelluna, Conegliano
  - Ospedale Umberto I, Mestre
  - Presidio Ospedaliero di Mirano, Mirano
  - Azienda Ospedaliera S. Maria, Terni
- Spain (6):
  - Complejo Hospitalario Arquitecto Marcide, Ferrol
  - Hospital Universitario de Madrid, Madrid
  - Hospital Montecelo, Mourente
  - Povisa, Salamanca
  - Hospital Clinico universitario de Santiago, Santiago de Compostela
  - Complejo Hospitalario Xeral-Cies, Vigo
- William Harvey Hospital, Ashford, United Kingdom